CLINICAL TRIAL: NCT03862014
Title: Clinical Evaluation of Permanent Molars With Molar Incisor Hypomineralization Treated With Silver Diamine Fluoride or Silver Modified Atraumatic Restorative Technique
Brief Title: Management of Molar Incisor Hypomineralization With Silver Diamine Fluoride or SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Zafer Cavit Cehreli, DDS, PhD, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: MIH-SDF/SMART
Record Dates: First submitted 2019-03-01; First posted 2019-03-05 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Dental Caries; Molar Incisor Hypomineralization
Keywords: molar incisor hypomineralization; silver diamine fluoride
MeSH Terms: conditions — Dental Caries; Molar Hypomineralization

STUDY DESIGN:
Intervention Model Description: Two materials on two molars in one patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SDF+KI (Experimental): SDF+KI will be applied on molars with MIH
  Interventions: Device: SDF+KI
- SMART(SDF+KI+GIC) (Active Comparator): SDF+KI+GIC will be applied on molars with MIH
  Interventions: Device: SDF+KI+GIC(SMART)

INTERVENTIONS:
Device: SDF+KI — Molar with MIH will be treated with SDF+KI
  Arms: SDF+KI
Device: SDF+KI+GIC(SMART) — Molar with MIH will be treated with SDF+KI+GIC(SMART)
  Arms: SMART(SDF+KI+GIC)

SUMMARY:
The purpose of this study is to evaluate and compare the clinical performance of Silver diamine Fluoride+Potassium Iodide (SDF+KI) and Silver-Modified Atraumatic Restorative Technique (SMART/SDF+KI+GIC) on molars with MIH

DETAILED DESCRIPTION:
SDF+KI and SMART (SDF+KI+GIC) were placed on two permanent molar teeth with MIH, in a split mouth design. 48 patients were included in the study. The teeth were randomized into two groups according to the dental restorative material.

Group 1: SDF+KI (Riva Star), Group 2: SDF+KI (Riva Star) +GIC (Equia Forte). The US Public Health Service criteria (secondary caries, anatomical form, marginal adaptation, marginal discoloration) was used for clinical evaluation of atraumatic resin restorations. The restorations were evaluated at baseline and 1., 6., 12., 18., 24. months. Intra-oral photos were taken directly after treatment and at control appointments to evaluate discoloration and seconder caries under magnification.

Fisher's Exact test, Kaplan-Meier Survival Curves, Log-rank test, Mann Whitney U test, and Friedman test was performed for the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients and parents of the patients who accept to participate and sign the informed consent
* Patients whose molar teeth are diagnosed as molar incisor hypomineralization by EAPD
* Teeth that are fully erupted
* Patients who have at least two permanent first molars that need fissure sealant
* Teeth that have white-yellow-brown discoloration that indicate high-caries risk

Exclusion Criteria:

* Teeth that are previously restored or have caries
* Patients who have orthodontic treatment
* Patients who are not cooperative for the dental procedure
* Teeth that have dental fluorosis or enamel malformation according to the specific syndromes

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Clinical performance of SDF+KI and SMART(SDF+KI+GIC) on molars with MIH | 2 years
  The US Public Health Service criteria (secondary caries, anatomical form, marginal adaptation, marginal discoloration) will be used for clinical evaluation of atraumatic resin restorations.

CONTACTS AND LOCATIONS:
Overall Officials: Zafer Cehreli, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
IPD is available from the corresponding author on reasonable request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 6 months after publication
Access Criteria: IPD is available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Erbas Unverdi G, Ballikaya E, Cehreli ZC. Clinical comparison of silver diamine fluoride (SDF) or silver-modified atraumatic restorative technique (SMART) on hypomineralised permanent molars with initial carious lesions: 3-year results of a prospective, randomised trial. J Dent. 2024 Aug;147:105098. doi: 10.1016/j.jdent.2024.105098. Epub 2024 May 24. PMID 38797490
- [Derived] Ballikaya E, Unverdi GE, Cehreli ZC. Management of initial carious lesions of hypomineralized molars (MIH) with silver diamine fluoride or silver-modified atraumatic restorative treatment (SMART): 1-year results of a prospective, randomized clinical trial. Clin Oral Investig. 2022 Feb;26(2):2197-2205. doi: 10.1007/s00784-021-04236-5. Epub 2021 Nov 6. PMID 34743243